CLINICAL TRIAL: NCT00842426
Title: A Pilot of Customized Continuous Care Management of Obesity in Pre-Diabetics
Brief Title: Evaluation of Lifestyle Interventions to Treat Elevated Cardiometabolic Risk in Primary Care
Acronym: E-LITE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Palo Alto Medical Foundation (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); American Heart Association (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, PhD, Associate Investigator, Palo Alto Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R34DK080878 (NIH)
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Obesity; Pre-diabetes; Metabolic Syndrome
Keywords: Diabetes; Cardiovascular disease; Metabolic syndrome; Cardiometabolic
MeSH Terms: conditions — Obesity; Glucose Intolerance; Metabolic Syndrome; Diabetes Mellitus; Cardiovascular Diseases | interventions — Self-Management

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Usual Care (No Intervention): Usual Care
- Self-Management Program (Experimental): Online Self-Management.
  Interventions: Behavioral: Self-management program (SM)
- Care Management Program (Experimental): Care management lifestyle modification program with intensive intervention phase with exercise and nutrition specialist. Followed by a online self-management phase.
  Interventions: Behavioral: Care management program (CM)

INTERVENTIONS:
Behavioral: Self-management program (SM) — Participants will attend a group orientation where the study nutritionist will provide an overview of the self-management lifestyle intervention program. Participants will receive instructions on how to use HeartHubTM, the American Heart Association's patient portal for information, tools, resources about cardiovascular risk assessment, goal setting, action planning, and self-monitoring.
  During the remainder of the 15-month intervention, participants will receive reminders on a regular basis to use the patient portal to assist in their ongoing self-management.
  Other Names: Self-monitoring and online tracking
  Arms: Self-Management Program
Behavioral: Care management program (CM) — In addition to participating in the activities described above, with the exception of the orientation session, participants in the Care Management Program will attend 12 weekly weight management classes during the initial 3 months. Classes will be co-led by a dietician and exercise specialist and will include a private weigh-in, a group discussion, a presentation of a lifestyle topic, 30 minutes of supervised moderate physical activity, followed by individual action-planning and goal-setting.
  During the remainder of the 15-month intervention, participants will continue to monitor their body weight, caloric intake, physical activity, and other data according to their care plan. In addition, study interventionist will follow up with participants regularly, via secure messaging or by phone, to provide ongoing counseling and support.
  Other Names: Intensive Lifestyle Program
  Arms: Care Management Program

SUMMARY:
The purpose of the E-LITE Study is to evaluate the feasibility and potential effectiveness of two lifestyle interventions in a community based primary care setting. The study aims to assess how changes in diet, exercise, and behavioral self-management affect weight and related risk factors for adults at risk for diabetes and cardiovascular disease.

DETAILED DESCRIPTION:
In the United States, there is an epidemic of obesity and, as a result, an epidemic of diabetes. Obese individuals with pre-diabetes (defined as impaired fasting glucose or impaired glucose tolerance) are at high risk for progression to diabetes. A vast majority of these individuals also have an increased risk of cardiovascular disease because of concomitant risk factors, such as abdominal obesity, dyslipidemia, and elevated blood pressure. Intensive lifestyle interventions that focus on dietary change, physical activity, and behavior modification have demonstrated efficacy in achieving and maintaining clinically significant (>5%) weight loss in populations of patients with pre-diabetes. However, the effectiveness, cost-effectiveness, generalizability, and sustainability of such interventions in routine primary care settings remain unknown, and rigorous clinical research is needed.

The primary hypothesis for the E-LITE Study is that the CM intervention will reduce BMI more than the SM intervention, which in turn will reduce BMI more than usual care, over 15 months. Secondarily, we hypothesize that, compared with usual care, intervention participants will be associated with greater improvements in waist circumference, lipids, blood pressure, blood glucose, lifestyle behaviors, and psychosocial well-being. In addition, we will examine the durability of weight loss and behavioral change in the months after the initial 3-month intensive stage.

ELIGIBILITY:
Inclusion Criteria:

* Ethnicity: All ethnic groups;
* Body mass index 25.0-39.9 kg/m2;
* Fasting plasma glucose between 100 and 125 mg/dL;
* Any two of the following: Waist circumference >40 inches in men, >35 inches in women (if in Asian American ≥ 35 inches in men; ≥31 inches in women); Triglycerides >150 mg/dL; High-density lipoprotein cholesterol (HDL-C) <40 mg/dL in men, <50 mg/dL in women; Systolic blood pressure >130 mm Hg or diastolic blood pressure >85 mm Hg.
* Having a primary care physician (PCP) at the PAMF Los Altos Center;
* Seen in primary or specialty care in the Palo Alto Region at least once in the preceding 24 months;
* A PAMF patient for ≥ 12 months;
* Able and willing to enroll and meet the requirements of the study.

Exclusion Criteria:

* Inability to speak, read or understand English;
* No regular access to a computer with Internet and email capabilities;
* Triglycerides >400 mg/dL;
* Systolic blood pressure >160 mm Hg or diastolic blood pressure >100 mm Hg;
* Initiation or change of drug therapy for elevated blood pressure or abnormal lipid levels within the past 3 months
* Having a medical (e.g., celiac disease) or social condition (e.g., religious beliefs) that precludes dietary changes;
* Having a medical or physical condition that make moderate intensity physical activity (like a brisk walk) difficult or unsafe;
* Use of weight-loss medications in the past 3 months;
* Regular use (> 5 days/month) of medications that affect appetite or weight (e.g., oral corticosteroids, insulin, certain oral hypoglycemics, certain antidepressants, etc.);
* Currently enrolled in a lifestyle intervention program at PAMF or elsewhere;
* Planning to undergo a bariatric surgery during the study period;
* Diagnosis of Type 1 or Type 2 diabetes mellitus;
* Significant medical co-morbidities, including uncontrolled metabolic disorders (e.g., thyroid, renal, liver), heart disease, stroke, and ongoing substance abuse;
* Renal insufficiency (i.e., GFR < 60 mL/min/1.73m2)
* Diagnosis of psychiatric disorders that would limit adequate informed consent or ability to comply with study protocol;
* Diagnosis of cancer (other than non-melanoma skin cancer) that was active or treated with radiation or chemotherapy within the past 2 years;
* Diagnosis of a terminal illness and/or in hospice care;
* Pregnant, lactating or planning to become pregnant during the study period;
* Already enrolled or planning to enroll in a research study that would limit full participation in this study or confound the observation and interpretation of the study's findings;
* Family/household member of another study participant or of a study staff member;
* No longer a PAMF patient or planning to transfer care outside of PAMF during the study period;
* Planning to move out of the area during the study period;
* PCP determination that the study is inappropriate or unsafe for the patient;
* Investigator discretion for clinical safety or protocol adherence reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2009-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | Baseline, 3-, 6- and 15- month follow-up

SECONDARY OUTCOMES:
Metabolic syndrome criterion factors: waist circumference, BP, FBG, TG, HDL, TG/HDL | Baseline, 6-, and 15-months
A1C, C-reactive protein | Baseline and 15-months
Dietary Intake | Baseline, 3-, 6-, and 15-months
Physical Activity | Baseline, 3-, 6-, and 15-months
Generic and Obesity-specific Health Related Quality of Life | Baseline, 3-, 6-, and 15-months
Patient and Physician Satisfaction | Baseline, 3-, 6-, and 15-months

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, M.D., Ph.D., Principal Investigator — Palo Alto Medical Foundation
Locations (1):
- Palo Alto Medical Foundation, Los Altos Center, Palo Alto, California, United States

REFERENCES:
- [Derived] Xiao L, Lv N, Rosas LG, Au D, Ma J. Validation of clinic weights from electronic health records against standardized weight measurements in weight loss trials. Obesity (Silver Spring). 2017 Feb;25(2):363-369. doi: 10.1002/oby.21737. Epub 2017 Jan 6. PMID 28059466
- [Derived] Azar KM, Xiao L, Ma J. Baseline obesity status modifies effectiveness of adapted diabetes prevention program lifestyle interventions for weight management in primary care. Biomed Res Int. 2013;2013:191209. doi: 10.1155/2013/191209. Epub 2013 Dec 4. PMID 24369008
- [Derived] Ma J, Yank V, Xiao L, Lavori PW, Wilson SR, Rosas LG, Stafford RS. Translating the Diabetes Prevention Program lifestyle intervention for weight loss into primary care: a randomized trial. JAMA Intern Med. 2013 Jan 28;173(2):113-21. doi: 10.1001/2013.jamainternmed.987. PMID 23229846
- [Derived] Yank V, Stafford RS, Rosas LG, Ma J. Baseline reach and adoption characteristics in a randomized controlled trial of two weight loss interventions translated into primary care: a structured report of real-world applicability. Contemp Clin Trials. 2013 Jan;34(1):126-35. doi: 10.1016/j.cct.2012.10.007. Epub 2012 Oct 31. PMID 23124047
- [Derived] Ma J, King AC, Wilson SR, Xiao L, Stafford RS. Evaluation of lifestyle interventions to treat elevated cardiometabolic risk in primary care (E-LITE): a randomized controlled trial. BMC Fam Pract. 2009 Nov 12;10:71. doi: 10.1186/1471-2296-10-71. PMID 19909549